CLINICAL TRIAL: NCT03530787
Title: Randomized Double-Blind Study of the Cosmetic Effects of Topical Acetyl Zingerone
Brief Title: Cosmetic Effects of Topical Acetyl Zingerone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1161176
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Wrinkle Appearance; Skin Pigment; Erythema; Side Effect; Microbiome; Lipidome
Keywords: Ginger; Curcumin; Zingerone
MeSH Terms: conditions — Pigmentation Disorders; Erythema | interventions — Floderm topical cream

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to two groups:
  AZ Group (n= 17) Control Group (n=17)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetyl Zingerone Group (Active Comparator): This group was given the topical with the active acetyl zingerone agent.
  Interventions: Other: Acetyl Zingerone Topical Cream
- Control Group (Placebo Comparator): This group was given the topical without the active acetyl zingerone agent and just the carrier lotion.
  Interventions: Other: Topical cream

INTERVENTIONS:
Other: Acetyl Zingerone Topical Cream — Topical cream with an active acetyl zingerone component.
  Other Names: Synoxyl AZ (Brand Name)
  Arms: Acetyl Zingerone Group
Other: Topical cream — Topical cream without an active acetyl zingerone component and just the carrier cream.
  Arms: Control Group

SUMMARY:
Cosmeceuticals are an emerging market within dermatology and the growth of natural products and derivatives of natural products has accelerated in use within the field. Here the investigators aimed to study the microbial and cosmetic effects of Synoxyl AZ, the trade name for topical acetyl zingerone (AZ), a novel compound designed based on Zingerone and curcumin.

DETAILED DESCRIPTION:
Cosmeceuticals are an emerging market within dermatology and the growth of natural products and derivatives of natural products has accelerated in use within the field. Here the investigators aim to study Synoxyl AZ, the trade name for topical acetyl zingerone (AZ), a novel compound designed based on Zingerone and curcumin.

Both curcumin and Zingerone are from the Zingiberacea family of plants (also known as the ginger family). Both have been widely studied and noted to have antibacterial effects and promote skin health effects. Curcumin has been studied widely in recent years due to various microbial effects. AZ is a derivative that is similar to both Zingerone and curcumin and has been noted to have many different activities including anti-inflammatory, antimicrobial, and antioxidant functions. However, there are no studies looking at how it modulates the skin cosmetically or the superficial microbiome.

The aim of this study was to compare the cosmetic effects of AZ to a vehicle over an 8-week period.

ELIGIBILITY:
Inclusion criteria:

* Individuals aged 30-60
* Healthy subjects

Exclusion Criteria:

* Those that have had topical antibiotics within the past 4 weeks
* Those that have had oral antibiotics within past 4 weeks
* Those who have used systemic isotretinoin in the last 6 months
* Those with a known allergy to members of the ginger family
* Current smokers OR 20 pack-year history of smoking OR Have smoked within the past 3 years
* Pregnant women
* Prisoners
* Those who have had any change to their hormonal birth control regimen in the last 4 weeks.
* Those with visible signs in the area of application of or on active treatment for cystic acne, eczema, seborrheic dermatitis, papulopustular rosacea at investigator discretion
* Those who have had a recent surgical or cosmetic procedure in the last 3 months that can affect facial wrinkles or facial hyperpigmentation, such as botulinum toxin injections, chemical peels, laser based therapies to the face, or face lift surgeries at investigator discretion

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Change in wrinkle appearance | 8 weeks
  Change in image based analysis of wrinkle severity from baseline
Change in appearance of skin pigmentation | 8 weeks
  Change in appearance of image based skin pigmentation from baseline

SECONDARY OUTCOMES:
Change in skin redness (erythema) | 4 weeks and 8 weeks
  Change in image based skin redness (erythema) and clinical assessment of redness from baseline
Change in appearance of skin pigmentation | 4 weeks
  Change in appearance of image based skin pigmentation from baseline
Change in wrinkle appearance | 4 weeks
  Change in image based analysis of wrinkle severity from baseline
Appearance of side effects such as scaling or irritation | 4 weeks and 8 weeks
  Appearance of side effects such as scaling or irritation from baseline
Change in superficial microbiome diversity | 4 weeks and 8 weeks
  Change in superficial microbiome diversity from baseline
Change in superficial lipidome diversity | 4 weeks and 8 weeks
  Change in superficial lipidome diversity from basline

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California-Davis, Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Semwal RB, Semwal DK, Combrinck S, Viljoen AM. Gingerols and shogaols: Important nutraceutical principles from ginger. Phytochemistry. 2015 Sep;117:554-568. doi: 10.1016/j.phytochem.2015.07.012. Epub 2015 Jul 27. PMID 26228533
- [Background] Vaughn AR, Haas KN, Burney W, Andersen E, Clark AK, Crawford R, Sivamani RK. Potential Role of Curcumin Against Biofilm-Producing Organisms on the Skin: A Review. Phytother Res. 2017 Dec;31(12):1807-1816. doi: 10.1002/ptr.5912. Epub 2017 Sep 7. PMID 28884496
- [Background] Vaughn AR, Branum A, Sivamani RK. Effects of Turmeric (Curcuma longa) on Skin Health: A Systematic Review of the Clinical Evidence. Phytother Res. 2016 Aug;30(8):1243-64. doi: 10.1002/ptr.5640. Epub 2016 May 23. PMID 27213821
- [Background] Ahmad B, Rehman MU, Amin I, Arif A, Rasool S, Bhat SA, Afzal I, Hussain I, Bilal S, Mir Mu. A Review on Pharmacological Properties of Zingerone (4-(4-Hydroxy-3-methoxyphenyl)-2-butanone). ScientificWorldJournal. 2015;2015:816364. doi: 10.1155/2015/816364. Epub 2015 May 27. PMID 26106644